CLINICAL TRIAL: NCT05334888
Title: Sex Hormone-specific Cardiovascular Risks in the Gut Microbiome-host Axis - A Longitudinal Cohort Study.
Brief Title: Sex-differential Host-microbiome CVD Risk - A Longitudinal Cohort Approach
Acronym: XCVD
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Dr. Lajos Marko, Dr., Charite University, Berlin, Germany
Other Study IDs: ChariteU - ECRC XCVD
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Transgender; Gut Microbiome; Immune System; Cardiovascular Risk Factors
Keywords: Transgender Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Sera Plasma Whole blood Feces Saliva Hair Skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The XCVD study investigates the influence of sex hormones on the composition of the gut microbiome and the possible emergence of cardiovascular risk factors. It will follow 200 healthy transgender individuals for two years during their hormone replacement therapy (HRT) and analyze them for the possible emergence of cardiovascular risk factors in relation to changes in the gut microbiome, metabolome, and immunome. We would also like to phenotype cardiovascular disease.

DETAILED DESCRIPTION:
Conducting this innovative study using established scientific methods such as omics platforms, systems biology, and careful CVD phenotyping will allow, for the first time, extensive data collection on the influence of sex hormones on the development of CVD risk factors as well as the role of the gut microbiome. In doing so, the influence of circulating sex hormones can also be quantified to potentially predict CVD risk markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Language requirements: German, English
* Previous gender hormone replacement therapy (HRT).
* Ability to give consent and written consent to participate.
* Health insurance (for clarification of incidental findings)

Exclusion Criteria:

* Diseases or functional disorders that, in the opinion of the study physician, preclude participation in the study.
* Incapacity or other circumstances that do not allow study participants to fully understand the nature, significance and scope of this study.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy transgender individuals during their gender hormone replacement therapy (HRT)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in relative species abundance of intestinal bacteria compared | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  baseline and 2 years after initiation of hormone replacement therapy. stool samples: Analysis with 16s rRNA sequencing

SECONDARY OUTCOMES:
Changes in cardio marker | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  sera: following cardio marker can be determined by Electro Chemiluminescence Immuno-Assay: BNP and hs-troponin.
Changes in hormone parameters | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  sera: following hormones can be determined by mass spectrometry: Free Androgen Index (fAI), Beta-CrossLaps (BCTX), Carboxy-terminal Propeptide of Procollagen I (P1CP), Luteinizing Hormone, Oestradiol, Progesterone, Testosterone, Free Testosterone, Sex Hormone Binding Globulin, Dihydrotestosterone, Oestron, Free Oestriol.
Changes in immune marker | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  sera: pro- and anti-inflammatory cytokines using cytokine - multiplex panel and Immune cell populations with shotgun sequencing
Changes in the concentration of of cortisol, progesterone, testosterone and dehydroepiandrosterone | Baseline, 2 years Follow Up
  Hair sample: Hair steroid analysis with Immunoassay and LC-MS/MS
Changes in the oral species abundance | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  saliva sample / oral / mouth: species abundance of oral bacteria (sequencing)
Changes in Immune cell marker / regulatory T-cells | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  Whole blood samples for Immune cell populations and peripheral blood mononuclear cells RNA isolation for whole-transcriptome shotgun sequencing.
Changes in Epigenomics | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  Whole blood samples for Immune cell populations and peripheral blood mononuclear cells RNA isolation for whole-transcriptome shotgun sequencing.
Changes in Proteomics | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  sera: MS and ELISA
Changes in Metabolomics | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  sera: MS and ELISA
Changes in relative species abundance of skin microbioma | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  skin swab: DNA - sequencing
Changes in BMI | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  body mass index (kg/m²)
Changes in circumference | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  circumference measurement (cm): waist and hip
Gender identity | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: Transgender Congruence Scale (TCS) & gender dysphoria
Changes in physical activity | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: International Physical Activity Questionnaire / IPAQ
Changes in mental health | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: Generalized Anxiety Disorder / GAD-7
Changes in Perceived Stress | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: Perceived Stress Questionnaire / PSQ
Changes in quality of life | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: quality of life / PROMIS
Changes in depression | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: Beck-Depressions-Inventar Revision / BDI II & The Patient Health Questionnaire (PHQ-9)
Changes in chrono type / sleep-wake behaviour | Baseline, 6, 12, 18 and 24 months Follow Up
  questionnaire: Munich ChronoType Questionnaire (MCTQ)
Changes in dietary habits | Baseline, 6, 12, 18 and 24 months Follow Up
  Food Frequency Quenstionnaire /FFQ, special diet and intake of dietary supplements, prebiotics and probiotics
Changes in socio-demographics | Baseline, 2 years Follow Up
  Family status, education level, current working status, and living situation
Documentation of HRT | Baseline - HRT start, 6, 12, 18 and 24 months Follow Up
  HRT medication, dosing, regimes, and progress as well as all transition -relevant surgery and physical changes
Changes in vital signs | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  Systolic and diastolic blood pressure and heart rate
Changes in life style risk parameters | Baseline, 2 years Follow Up
  Smoking status, alcohol consumption and use of recreational drugs
Changes in CVD risk scores | Baseline, 2 years Follow Up (optional: after 1 year Follow Up)
  Framingham risk scores (FRS) and Systematic Coronary Risk Evaluation (SCORE)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Forslund, Dr., Study Director — Max-Delbrück-Center; Lajos Marko, Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Experimental and Clinical Research Center, Clinical Research Unit, Berlin, Germany

REFERENCES:
- [Result] Fromentin S, Forslund SK, Chechi K, Aron-Wisnewsky J, Chakaroun R, Nielsen T, Tremaroli V, Ji B, Prifti E, Myridakis A, Chilloux J, Andrikopoulos P, Fan Y, Olanipekun MT, Alves R, Adiouch S, Bar N, Talmor-Barkan Y, Belda E, Caesar R, Coelho LP, Falony G, Fellahi S, Galan P, Galleron N, Helft G, Hoyles L, Isnard R, Le Chatelier E, Julienne H, Olsson L, Pedersen HK, Pons N, Quinquis B, Rouault C, Roume H, Salem JE, Schmidt TSB, Vieira-Silva S, Li P, Zimmermann-Kogadeeva M, Lewinter C, Sondertoft NB, Hansen TH, Gauguier D, Gotze JP, Kober L, Kornowski R, Vestergaard H, Hansen T, Zucker JD, Hercberg S, Letunic I, Backhed F, Oppert JM, Nielsen J, Raes J, Bork P, Stumvoll M, Segal E, Clement K, Dumas ME, Ehrlich SD, Pedersen O. Microbiome and metabolome features of the cardiometabolic disease spectrum. Nat Med. 2022 Feb;28(2):303-314. doi: 10.1038/s41591-022-01688-4. Epub 2022 Feb 17. PMID 35177860
- [Result] Talmor-Barkan Y, Bar N, Shaul AA, Shahaf N, Godneva A, Bussi Y, Lotan-Pompan M, Weinberger A, Shechter A, Chezar-Azerrad C, Arow Z, Hammer Y, Chechi K, Forslund SK, Fromentin S, Dumas ME, Ehrlich SD, Pedersen O, Kornowski R, Segal E. Metabolomic and microbiome profiling reveals personalized risk factors for coronary artery disease. Nat Med. 2022 Feb;28(2):295-302. doi: 10.1038/s41591-022-01686-6. Epub 2022 Feb 17. PMID 35177859
- [Derived] Franz K, Marko L, Mahler A, Chakaroun R, Heinitz S, Schlogl H, Sacher J, Steckhan N, Dechend R, Adams N, Andersen M, Glintborg D, Viehweger M, Bahr LS, Forslund-Startceva SK. Sex hormone-dependent host-microbiome interactions and cardiovascular risk (XCVD): design of a longitudinal multi-omics cohort study. BMJ Open. 2025 Jan 9;15(1):e087982. doi: 10.1136/bmjopen-2024-087982. PMID 39788783
- See also: Short proposal of the study — https://www.mdc-berlin.de/de/forslund